CLINICAL TRIAL: NCT04855292
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Dose Phase Ib Study in Overweight/Obese Subjects Without Diabetes to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of TG103 Injection
Brief Title: A Study of TG103 Injection in Overweight/Obese Subjects Without Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSA1803-CSP-004
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TG103 injection 15 mg (Experimental): TG103 injection (15 mg, N=12) and Placebo (N=4) will be administered subcutaneously once weekly in overweight/obese non-diabetic subjects.
  Interventions: Drug: TG103 injection; Drug: Placebo
- TG103 injection 22.5 mg (Experimental): TG103 injection (22.5 mg, N=12) and Placebo (N=4) will be administered subcutaneously once weekly in overweight/obese non-diabetic subjects.
  Interventions: Drug: TG103 injection; Drug: Placebo
- TG103 injection 30 mg (Experimental): TG103 injection (30 mg, N=12) and Placebo (N=4) will be administered subcutaneously once weekly in overweight/obese non-diabetic subjects.
  Interventions: Drug: TG103 injection; Drug: Placebo

INTERVENTIONS:
Drug: TG103 injection — TG103 injection, SC, once weekly
Drug: Placebo — Placebo control, SC, once weekly

SUMMARY:
The main purpose of this study is to assess the safety and tolerability of multiple doses of TG103 injection in overweight/obese subjects without diabetes

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, multiple-doses, parallel-group study to characterize the safety (including the anti-drug antibodies (ADA)), tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of TG103 injection. The study will consist of 3 periods: an approximately 4-week screening period, followed by a 12-week treatment period, and a 3-week safety follow-up period. Eligible subjects will be enrolled into three paralleled dose groups (15 mg, 22.5 mg and 30 mg) with 16 subjects in each group. Within each group, subjects will be randomized in a 3:1 ratio to receive TG103 injection or placebo subcutaneously (SC) once a week (QW) over a period of 12 weeks. Each group will be started at a low dose of 7.5 mg and gradually up-titrated at weekly intervals until the target dose.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years (inclusive); no gender limitation;
2. Body mass index (BMI) ≥ 26.0 kg/m2, BMI = weight(kg)/height2 (m2); body weight ≥ 60 kg; Stable body weight (less than 5% self-reported change within 3 months);
3. Fasting blood glucose 3.9-7.0 mmol/L (exclusive) and the HbA1c < 6.5%;
4. Subjects of childbearing age must use reliable methods of contraception from the date of signing an informed consent to at least 6 months after the last dose;
5. Subjects who fully understand the study, voluntarily participate in the trial and sign the informed consent form。

Exclusion Criteria:

1. History of allergy to Glucagon-like peptide-1 (GLP-1) analogues, or history of serious allergy to drugs or food;
2. Secondary obesity, such as obesity induced by metabolic disease (e.g., Cushing's syndrome, hypothyroidism etc.) or drug treatment (e.g. with corticosteroids, tricyclic anti-depressants, atypical anti-psychotics);
3. Subjects have confirmed diagnosis of type 1 or type 2 diabetes;
4. History of or current pancreatitis (history of chronic or acute pancreatitis);
5. Previous clinically significant abnormal gastric emptying (e.g., gastric outlet obstruction) and severe chronic gastrointestinal diseases (e.g., active ulcer within 6 months);
6. Individual or family history of medullary thyroid cancer (MTC), type 2 multiple endocrine neoplasia syndrome or other hereditary diseases predisposing to MTC; abnormal and clinically significant thyroid function at screening, requiring pharmacological treatment or not yet clinically stable after treatment;
7. Subjects with history of or current cholestasis or gallbladder stones (previous gallstone removal or lithotripsy) and/or cholecystectomy, who have no further sequelae, can enter into the study at the discretion of the investigator after assessing the risk;
8. History of chronic malabsorption syndrome;
9. Subjects with hematological diseases (e.g., aplastic anemia, myelodysplastic syndrome) or any disease causing hemolysis or erythrocyte instability (e.g., malaria);
10. Severe systemic infectious diseases within 1 month prior to screening;
11. Systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg during screening;
12. Any of the following serious cardiovascular and cerebrovascular events prior to screening: unstable angina pectoris requiring hospitalization, myocardial infarction, coronary artery bypass grafting, percutaneous coronary intervention (except for diagnostic angiography), moderate to severe congestive heart failure (NYHA grade III or IV), atrial or ventricular arrhythmia requiring hospitalization (e.g., atrial fibrillation, ventricular tachycardia, tec.), second degree or third degree atrioventricular block without a pacemaker, clinically significant long QT syndrome or prolonged QTc interval, signs of localized ischemic heart disease, pacemaker or defibrillator implantation, stroke or transient ischemic attack or cerebrovascular accident within 6 months, or planned coronary artery bypass grafting or revascularization;
13. The white blood cell count exceeds 10% of the normal range, or hemoglobin<100 g/L during the screening period;
14. Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≥ 2.5 x upper limit of normal (ULN), or fasting triglyceride ≥ 5.64 mmol/L or eGFR < 60mL/(min*1.73 m2) during the screening period;
15. History of severe respiratory tract, blood system, central nervous system diseases (e.g., epilepsy, etc.), or history of malignant tumor, mental diseases (e.g., depression, anxiety, etc.), or history of other diseases that may endanger the safety of the subjects and are considered unsuitable for this study in the investigator's opinion;
16. Use of approved weight-lowering pharmacotherapy (e.g., orlistat) within 3 months prior to the first dose;
17. History of surgical treatment for obesity (except for liposuction performed one year ago);
18. Have used incretin analogues or other drugs that might interfere with the trial in the opinion of the investigator within 3 months before the first dose;
19. History of drug abuse or dependence within 5 years prior to screening, with a positive urine drugs of abuse testing at screening;
20. Average alcohol intake is more than 21 units of alcohol (male)/14 units of alcohol (female) per week within the 3 months prior to screening, or positive alcohol breath test before administration;
21. Smoke more than 5 cigarettes per day within 3 months prior to screening;
22. Blood lost ≥ 400 mL due to trauma or major surgery or blood donation ≥ 400 mL within 3 months prior to screening;
23. Have participated in any clinical trial involving an investigational product within 3 months prior to screening;
24. Vaccinated within 28 days before screening or planned to be vaccinated within 1 week after receiving the study drug;
25. Have a positive test result for hepatitis B surface antigen, hepatitis C antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
26. Pregnant (blood pregnancy test positive at screening) and lactating female, or male and female planned to have children during the trial or within 6 months after the last dose;
27. Not suitable for this study in the investigator's opinion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by incidence and severity of adverse events | Up to 99 days

SECONDARY OUTCOMES:
PK profile-AUC: Area under the plasma concentration versus time curve | Day1, 8, 15, 22, 29, 64, 71, and 78
PK profile- Cmax: Peak Plasma Concentration | Day1, 8, 15, 22, 29, 64, 71, and 78
PK profile- Tmax: Time to maximum plasma concentration | Day1, 8, 15, 22, 29, 64, 71, and 78
PK profile- t1/2: Half time | Day1, 8, 15, 22, 29, 64, 71, and 78
PK profile- CL/F: Apparent clearance | Day1, 8, 15, 22, 29, 64, 71, and 78
PD profile- Weight change relative to baseline | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85 and 99
PD profile- Proportion of subjects with a baseline weight loss of more than 5 percent | Day1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, 85 and 99
PD profile- Waistline change relative to baseline | Day8, 15, 22, 29, 43, 57, 71, 78, 85 and 99
PD profile- Change of waist-hip ratio relative to baseline | Day8, 15, 22, 29, 43, 57, 71, 78, 85 and 99
PD profile- Change of blood pressure（systolic blood pressure and diastolic blood pressure）relative to baseline | Day15, 22, 29, 43, 85 and 99
PD profile- Change of blood fat levels relative to baseline | Day15, 22, 29, 43, 85 and 99
The occurrence of TG103 anti-drug antibodies (ADA) | Day1, 15, 29, 57, and 99

CONTACTS AND LOCATIONS:
Locations (1):
- Gao Huanhuan, Beijingcun, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin D, Xiao H, Yang K, Li J, Ye S, Liu Y, Jing S, Lin Y, Yang Y, Huang L, Yuan J, Li Z, Yang J, Gao H, Xie Y, Xu M, Yan L. Safety, tolerability, pharmacokinetics, and pharmacodynamics of TG103 injection in participants who are overweight or obese: a randomized, double-blind, placebo-controlled, multiple-dose phase 1b study. BMC Med. 2024 May 29;22(1):209. doi: 10.1186/s12916-024-03394-z. PMID 38807146